CLINICAL TRIAL: NCT00410722
Title: Effect of Nuts on Glycemic Control and Cardiovascular Disease Risk in Type 2 Diabetes
Brief Title: Effect of Nuts vs. a Wheat Bran Muffin in Type 2 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, David Jenkins, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 06-274
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes; Cardiovascular Disease; Diet Therapy
Keywords: Nutrition; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Full-Dose Nut (Experimental): Subjects will be given tree nuts (almonds, hazelnuts, pistachios, macadamia nuts, pecans, walnuts, and cashews) and peanuts (at a predetermined amount to consume based on their recommended energy intake), and advised to follow a diabetic diet.
  Interventions: Dietary Supplement: Mixed tree nuts
- Half-Dose Nut (Experimental): Subjects will be given tree nuts (almonds, hazelnuts, pistachios, macadamia nuts, pecans, walnuts, and cashews) and peanuts as well as the control supplement (wheat bran muffin)(at a predetermined amount to consume based on their recommended energy intake), and advised to follow a diabetic diet.
  Interventions: Dietary Supplement: Whole wheat and bran muffin; Dietary Supplement: Mixed tree nuts
- Control (Active Comparator): Subjects will be given a control supplement (wheat bran muffin)(at a predetermined amount to consume based on their recommended energy intake), and advised to follow a diabetic diet.
  Interventions: Dietary Supplement: Whole wheat and bran muffin

INTERVENTIONS:
Dietary Supplement: Whole wheat and bran muffin
  Arms: Control; Half-Dose Nut
Dietary Supplement: Mixed tree nuts
  Arms: Full-Dose Nut; Half-Dose Nut

SUMMARY:
To determine if tree nuts (Almonds, Hazelnuts, Pistachios, Peanuts, Macadamia nuts, Pecans, Walnuts and Cashews) improve glycemic control in type 2 diabetes, as assessed by HbA1c and serum fructosamine, and to assess whether these outcomes relate to improvements in cardiovascular health (i.e. plasma lipids and measures of oxidative stress, inflammatory biomarkers and nitric oxide generation). The investigators have found that nuts tend to reduce the glycemic index of bread and have little effect of raising blood glucose on their own. Therefore the investigators believe that they would be ideal foods to displace high glycemic foods from the diet and lower the dietary glycemic load. This will result in improved blood glucose control in type 2 diabetes, with additional benefits on coronary heart disease risk factors due to other effects of nuts.

DETAILED DESCRIPTION:
The investigators wish to study the effect of nuts on glycemic control and to confirm their lipid lowering effects in type 2 diabetes. The consumption of nuts with their high unsaturated fat, vegetable protein (arginine) and fiber contents will decrease the glycemic load of the diet and improve glycemic control. The investigators anticipate that the favorable fatty acid profile of nuts along with the vegetable protein will improve the blood lipid profile in type 2 diabetes and thereby establish a cardiovascular risk reduction associated with nuts in this population.

Furthermore, flavonoids and vitamin E present in high concentrations in nuts, and known to have antioxidant activity may help to counter the elevated oxidative stress and inflammation experienced by diabetics. The investigators will therefore determine the effect of nut feeding on measures of oxidative stress (including oxidized low-density lipoprotein cholesterol (LDL-C), considered to be of direct relevance to coronary heart disease), inflammation (C-reactive protein, serum amyloid A and interleukin-6) and nitric oxide metabolism (blood nitric oxide and nitrotyrosine levels). These data would further add to interest in nuts in relation to cardiovascular disease risk reduction and diabetic complications.

Background Diet: A diet conforming to the American Diabetes Association (ADA) and National Cholesterol Education Program (NCEP) Adult Treatment Panel III guidelines. Nuts, soy and dietary supplements (vitamins, minerals, herbal remedies) will be excluded in the background diet during all phases of the study.

Treatment diets:(1) Full-Dose Nut Diet: Raw nuts will be added as supplements to the subject's usual diet. Subjects with calorie needs of 2,400 kcal or greater, assessed by Lipid Research Clinic (LRC) tables, will receive the full-dose supplement (100 g/d of nuts, approximately 600 kcal). Subjects requiring between 1,600-2,400 kcal daily will receive 75% of the full-dose supplement (75 g/d of nuts, approximately 450 kcal). Subjects requiring less than 1,600 kcal daily will receive 50% of the full-dose supplement (50 g/d of nuts, approximately 300 kcal). (2) Half-Dose Nut Diet: Raw nuts will be added as supplements to the subject's usual diet. Subjects with calorie needs of 2,400 kcal or greater, assessed by LRC tables, will receive half of the full dose of the nut supplement (50 g/d of nuts, approximately 300 kcal) with the rest of the calories provided by the muffin (2 muffins are 300 kcal) for a total of 600 kcal. Subjects requiring between 1,600-2,400 kcal daily will receive 75% of the half-dose supplement (37.5 g/d of nuts and 1.5 muffins, approximately 450 kcal). Subjects requiring less than 1,600 kcal daily will receive 50% of the half-dose supplement (25 g/d of nuts and 1 muffin, approximately 300 kcal). (3): The full-dose control supplement will be four 150 kcal muffins. Control supplements will be matched with the energy content of the nut supplements, i.e. either 600 kcal/d (4 muffins); 450 kcal/d (3 muffins); 300 kcal/d (2 muffins). The macronutrient composition of the muffins will conform to an NCEP Step 2 diet with 25% total fat, <7% saturated fat by use of corn oil as the oil commonly used in healthy baked goods, with 18% protein (the average for our subject population) using added skim milk powder, and zero cholesterol. Muffins will be made with whole wheat flour.

Diet History: one-week weighed diet histories will be obtained prior to the start and at weeks 4, 8 and 12 of the study for assessment of macronutrients, dietary fiber and fatty acids.

Palatability/Satiety: for palatability and satiety, subjects will record their ratings using a 7-point bipolar semantic scale at monthly intervals during each study phase.

Anthropometry and Blood Pressure: height at recruitment and body weight, blood pressure, waist and hip circumference, and body composition will be taken immediately prior to and at each clinic visit (wk 0, 2, 4, 8, 10, 12) during the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and post menopausal women with type 2 diabetes treated with diet plus oral hypoglycemic agents (sulfonylureas (glyburide), biguanides (metformin), Thiazolidinediones (TZDs) and new secretagogues (Repaglinide)) at a stable dose for at least 3 months prior to starting the study;
* HbA1c of 6.5 to 8.0% as a compromise between those whose levels are acceptable and the level which is currently considered unacceptable.
* Diabetes diagnosed >6 months prior to randomization
* Weight stable within 3% body weight >2 months.

Exclusion Criteria:

* Use of acarbose
* Use of Insulin
* Known nut allergies
* Clinically significant gastroparesis
* Use of steroids
* Presence of GI disease (celiac disease, ulcerative colitis, and Crohns)
* Major cardiovascular event (stroke or myocardial infarction)
* Major surgery < 6 months prior to randomization
* Presence of major debilitating disorder such as clinically significant liver disease (not including non-alcoholic fatty liver (NAFL) or non-alcoholic steatohepatitis (NASH) but including cirrhosis, infectious hepatitis (B and C), aspartate transaminase (AST) or alanine transaminase (ALT) > 130 IU/L)
* Renal failure (high creatinine > 150 mmol/L)
* Serum triglyceride > 6 mmol/L.
* Patients currently undergoing treatment for cancer with the exception of non-melanoma skin cancer, but not high risk patients or those whose treatment has been successfully completed.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Markers of glycemic control: Fasting serum fructosamine | From prestudy and week 0, to end of treatment weeks 8, 10, 12
Fasting serum HbA1c | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
Fasting glucose | From prestudy and week 0, to end of treatment and weeks 8, 10, and 12
Fasting insulin | From prestudy and week 0, to end of treatment and weeks 8, 10, and 12

SECONDARY OUTCOMES:
24h urinary C-peptide excretion | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
Branched chain amino acids | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
Serum triglyceride | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
Very Low-Density Lipoprotein (VLDL) triglyceride | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
VLDL-C | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
LDL:HDL-C | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
Apolipoprotein B:A1 | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
Lipoprotein(a) | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
oxidized LDL | From beginning of study, week 0, to end of treatment week 12
markers of oxidative stress | From beginning of study, week 0, to end of treatment week 12
C-reactive protein | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
markers of inflammation | From prestudy and week 0, to end of treatment weeks 8, 10, and 12
Cancer cell proliferation | From beginning of study, week 0, to end of treatment week 12

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, MD, PhD, Principal Investigator — University of Toronto, St. Michael's Hospital; Cyril WC Kendall, PhD, Study Chair — University of Toronto, St. Michael's Hospital
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jenkins DJA, Kendall CWC, Lamarche B, Banach MS, Srichaikul K, Vidgen E, Mitchell S, Parker T, Nishi S, Bashyam B, de Souza RJ, Ireland C, Pichika SC, Beyene J, Sievenpiper JL, Josse RG. Nuts as a replacement for carbohydrates in the diabetic diet: a reanalysis of a randomised controlled trial. Diabetologia. 2018 Aug;61(8):1734-1747. doi: 10.1007/s00125-018-4628-9. Epub 2018 May 23. PMID 29789878
- [Derived] Nishi SK, Kendall CW, Bazinet RP, Bashyam B, Ireland CA, Augustin LS, Blanco Mejia S, Sievenpiper JL, Jenkins DJ. Nut consumption, serum fatty acid profile and estimated coronary heart disease risk in type 2 diabetes. Nutr Metab Cardiovasc Dis. 2014 Aug;24(8):845-52. doi: 10.1016/j.numecd.2014.04.001. Epub 2014 May 13. PMID 24925120
- [Derived] Jenkins DJ, Kendall CW, Banach MS, Srichaikul K, Vidgen E, Mitchell S, Parker T, Nishi S, Bashyam B, de Souza R, Ireland C, Josse RG. Nuts as a replacement for carbohydrates in the diabetic diet. Diabetes Care. 2011 Aug;34(8):1706-11. doi: 10.2337/dc11-0338. Epub 2011 Jun 29. PMID 21715526 (Retraction: PMID 26798151 Diabetes Care. 2016 Feb;39(2):319)